CLINICAL TRIAL: NCT03346278
Title: Text Messaging to Improve Heart Healthy Behaviors and Cardiac Rehabilitation Participation
Brief Title: Text Message Intervention to Improve Cardiac Rehab Participation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator leaving institution. 38 subjects were enrolled in Aim 1. Aim 2 was not initiated.
Sponsor: University of Washington (Other)
Collaborators: John L. Locke Jr. Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Alexis Beatty, Assistant Professor, Department of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003125
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention; Coronary Artery Bypass Surgery; Heart Valve Repair or Replacement; Heart Transplant; Left Ventricular Assist Device; Chronic Stable Angina; Chronic Stable Heart Failure
Keywords: Cardiac Rehabilitation; Text Messaging
MeSH Terms: conditions — Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Text Message Intervention (No Intervention): Participants will receive usual care of information on CR and clinical referral to CR.
- Text Message Intervention (Experimental): Participants randomized to the intervention will receive usual care plus a text messaging intervention.
  Interventions: Behavioral: Text Messaging Intervention

INTERVENTIONS:
Behavioral: Text Messaging Intervention — After completing baseline procedures, study staff will activate the intervention in the participant's profile on the text messaging platform if the participant was randomized to the intervention. The text messaging platform will deliver messages by an automated algorithm. Participants will receive 4 messages per week for 6 months.
  Arms: Text Message Intervention

SUMMARY:
Cardiac rehabilitation (CR) is strongly recommended for patients with coronary heart disease. However, patient enrollment and completion of cardiac rehabilitation is low. This study will examine if a mobile phone intervention that uses a text messaging program can successfully promote participation in cardiac rehabilitation.

DETAILED DESCRIPTION:
Mobile phone interventions, such as text messaging programs, have been shown to promote healthy behaviors in patients with coronary heart disease, but it is unknown whether text messaging can successfully promote participation in cardiac rehabilitation.

This study will have the following aims:

Aim 1: Adapt a theory- and evidence-based text messaging intervention to promote participation in cardiac rehabilitation.

Aim 2: Determine whether text messaging improves participation in cardiac rehabilitation among eligible patients.

This study will have two parts. In part 1, the investigators will enroll patients with heart disease to rate the acceptability of text messages. In part 2, the investigators will enroll patients to participate in a randomized controlled trial. Participants will be randomized to receive text messages or no text messages for 6 months. Those who have been assigned to receive the text messaging intervention will be sent several text messages per week throughout the study period. The content of these text messages is designed promote healthy behaviors and participation in cardiac rehabilitation. Those who have not been assigned to receive the text messaging intervention will receive usual care. Outcome measures will be assessed at a baseline visit and at a 6-month follow-up visit at the end of the intervention. Additionally, some participants in the text messaging intervention group will be interviewed about their overall satisfaction and engagement with the text messages upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Diagnosis eligible for cardiac rehabilitation within 90 days (myocardial infarction, percutaneous coronary intervention, coronary artery bypass surgery, heart valve repair/replacement, heart transplant, left ventricular assist device, chronic stable angina, chronic stable heart failure)
* Part 2: Hospitalized for diagnosis eligible for cardiac rehabilitation (myocardial infarction, percutaneous coronary intervention, coronary artery bypass surgery, heart valve repair/replacement, heart transplant, left ventricular assist device)
* Eligible for cardiac rehabilitation
* Owns a smartphone capable of receiving and sending SMS text messages

Exclusion Criteria:

* Unable to communicate in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Attendance at cardiac rehab | 6 months
  Documented attendance at one or more cardiac rehab sessions. Primary analysis will compare the proportion attending cardiac rehab in the text message intervention and no text message intervention arms.

SECONDARY OUTCOMES:
Number of cardiac rehab sessions attended | 6 months
  Documented attendance at cardiac rehab sessions
Physical activity | 6 months
  Self-reported via International Physical Activity Questionnaire (IPAQ) - Total physical activity in continuous MET-min/week. Total physical activity is the sum of walking, moderate, and vigorous physical activity. Walking MET-minutes/week = 3.3 * walking minutes * walking days. Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days. Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days.
Exercise capacity | 6 months
  6-minute walk test (6MWT)
Tobacco use | 6 months
  Participant self-report of tobacco use in past 30 days
Diet | 6 months
  Self-reported diet via Rate Your Plate questionnaire. Score 23-69, with 69 representing best diet.
Blood pressure | 6 months
  Blood pressure measured by study staff
Body Mass Index (BMI) | 6 months
  Weight measured by study staff. BMI = weight (kg) / height in meters squared (m2)
Cholesterol (LDL) | 6 months
  Obtained from medical records
Disease-specific health status | 6 months
  Self-reported health status via validated Seattle Angina Questionnaire (SAQ) - Short Form for participants with ischemic heart disease. The questionnaire is scored from 0-100 with 100 being the highest reportable health status. SAQ domains will include: Physical Limitation, Angina Frequency, and Quality of Life.
Disease-specific health status | 6 months
  Self-reported health status via validated Kansas City Cardiomyopathy Questionnaire (KCCQ) - Short Form for participants with heart failure or valvular heart disease. The questionnaire is scored from 0-100 with 100 being the highest reportable health status. KCCQ domains will include: Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitation.
Depressive symptoms | 6 months
  Self-reported depressive symptoms via Patient Health Questionnaire-9 (PHQ-9). Scored 0-27 with 0 representing no depressive symptoms and 27 representing severe depressive symptoms.
Patient activation | 6 months
  Self-reported activation via the Patient Activation Measure 13 (PAM-13)
Patient satisfaction | 6 months
  Self-reported satisfaction with the intervention
Patient experience | 6 months
  Self-reported experience with the intervention
Hospitalizations | 6 months
  Confirm participant-reported events from medical records. We will report a composite of number of participants with Hospitalizations, ER visits, or Death, as well as number of participants with each individual outcome.
ER visits | 6 months
  Confirm participant-reported events from medical records. We will report a composite of number of participants with Hospitalizations, ER visits, or Death, as well as number of participants with each individual outcome.
Death | 6 months
  Confirm participant-reported events from medical records. We will report a composite of number of participants with Hospitalizations, ER visits, or Death, as well as number of participants with each individual outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Beatty, MD, MAS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share via University of Washington research data repository after the conclusion of the study and publication of findings